CLINICAL TRIAL: NCT05927467
Title: Study of the Natural History of Alport Syndrome by Establishment of an International Database
Brief Title: Eurbio-Alport (RaDiCo Cohort) (RaDiCo Eurbio-Alport)
Acronym: Eurbio-Alport
Status: Recruiting | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-82
Record Dates: First submitted 2021-12-20; First posted 2023-07-03 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Alport Syndrome
Keywords: Alport Syndrome; Rare disease; European database; Quality of life; Kidney disease; Molecular diagnostics; Predictive biomarkers
MeSH Terms: conditions — Nephritis, Hereditary; Rare Diseases; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Alport syndrome is a rare, inherited condition characterized by a combination of glomerular nephropathy progressing to kidney failure, deafness, and eye involvement. This disease is associated with mutations in the genes encoding one of the three IV collagen chains expressed in the glomerular basement membrane. Significant progress has been made in understanding the molecular mechanisms responsible for the disease, but relatively little in understanding the progression of renal failure and in the area of therapeutics. We have shown in a retrospective European study that blockers of the renin angiotensin system may slow disease progression, but no controlled studies have been performed. Finally, innovative therapies (anti-micro-RNA, stem cells) have recently shown their effectiveness in animal models of the disease, and industrials are planning to quickly carry out phase 1 trials to test molecules. Carrying out therapeutic trials in humans will require full knowledge of the natural history of the disease (isolated hematuria, microalbuminuria, macroalbuminuria, renal failure and its progression) and gathering a sufficient number of patients, especially in the early stages. These trials and the indications for treatments would be greatly facilitated by the discovery of biomarkers that make it possible to predict the progression to renal failure earlier than the onset of proteinuria.

The study aims to:

* Establish a European database on Alport syndrome to assess the natural history of the disease.
* To investigate the impact of the disease on the educational and professional life of patients and their families, and on the adherence and tolerance to renin-angiotensin system blockers prescribed to proteinuric patients.
* Investigate access to molecular diagnostics and genetic counseling, as well as identify biomarkers that can predict progression of kidney disease.

This project will be carried out at a French level with the support and participation of the very active renal rare disease sector, in collaboration with various countries wishing to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AS based on electron microscopic examination of the renal biopsy and/or molecular studies and/or abnormal expression of type IV collagen chains on skin and/or glomerular basement membranes.
* Signed informed consent

Exclusion Criteria:

- No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The countries that are potentially interested in joining the project have identified in their local records about 100 (Germany), 200 (Spain), 100 (United Kingdom), 785 (Italy), 100 (Belgium) patients. The database ASTOR in USA have included 800 patients. For France, the CEMARA database contains currently 680 Alport Syndrome patients while there are 950 identified patients in France. These patients are followed in nephrology and paediatric nephrology services belonging to the French network for rare renal diseases. Prevalent cases will include cases already registered in the different existing databases in the different countries, after monitoring that the inclusion criteria are respected. There is no known estimated incident rate, but according to the available information and the estimated prevalence rate (1/5,000), it is expected to enrol roughly between 100 and 200 incident patients/year in the study.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2017-05-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Renal function: eGFR, age at ESRD, requirement of Renal Replacement Therapy (RRT) and type of RRT | Through study completion, at 1 year, 2 year, 3 year
Urine bio-analysis results: Presence or not and quantification of hematuria, microalbuminuria and proteinuria | Through study completion, at 1 year, 2 year, 3 year
Presence or not of hypertension | Through study completion, at 1 year, 2 year, 3 year
Level of Hearing loss | Through study completion, at 1 year, 2 year, 3 year
Ocular symptoms (presence or not of lenticonus, cataract, retina and cornea impairment) | Through study completion, at 1 year, 2 year, 3 year

SECONDARY OUTCOMES:
Adverse events for the long-term safety of RAAS blockers treatment | Through study completion, at 1 year, 2 year, 3 year
Quality of life questionnaires | Through study completion, at 1 year, 2 year, 3 year
  Impact of disease on quality of life will be evaluated through scores of quality of life questionnaires SF36 for Adult et SF10 for paediatric patients
Compliance | Throughout the follow-up
  Compliance will be evaluated using X. Girerd Compliance Questionnaire

OTHER OUTCOMES:
Disease stage | Throughout the follow-up
  Stratification of patients according to their disease stage; patients' distribution analysis among countries
Urinal concentration of specific molecules | Through study completion, at 1 year, 2 year, 3 year
  Correlation assessment between the urinal concentration of the five molecules recently described by Terzi's lab as predicting progression of CKD (or other putative biomarkers) with the rate of decline of the GFR (according of the estimated GFR) on a 3 year- period

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Heidet, PHD, Principal Investigator — INSERM U933
Locations (1):
- RaDiCo Eurbio-Alport, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided